CLINICAL TRIAL: NCT03970226
Title: A Phase 0/Feasibility Trial of Tocilizumab in Children and Adolescents With Newly- Diagnosed or Recurrent/Progressive Adamantinomatous Craniopharyngioma
Brief Title: Tocilizumab in Children With ACP
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2143.cc; R03CA235200 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-05-31 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Adamantinomatous Craniopharyngioma
Keywords: Phase 0; Feasibility; Tocilizumab
MeSH Terms: conditions — Craniopharyngioma | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Phase 0 to open first and if outcomes are favorable showing drug penetration then the Feasibility Phase will open. Both arms will be open concurrently.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab Administration: Phase 0 (Experimental): In Phase 0, patients will receive one dose of tocilizumab prior to surgery.
  Interventions: Drug: Tocilizumab
- Tocilizumab Administration: Feasibility Phase (Experimental): During the Feasibility Phase, patients will receive tocilizumab every 2 weeks for up to 13 cycles (approximately 1 year). Patients will be followed for up to 5 years.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Phase 0: One dose of tocilizumab prior to surgery
  Feasibility phase: Tocilizumab administered every 2 weeks for up to 13 cycles (approximately 1 year).
  Other Names: Actemra

SUMMARY:
This study will be conducted in two phases. The first phase (phase 0) will be looking at patients with new or recurrent/ progressed craniopharyngioma tumors. These patients will be given one dose of tocilizumab before they have SOC surgery of their tumor. The objective of this phase is to see if drug reaches the tumor. If phase 0 is favorable and shows that drug is penetrating the tumor, the second phase of the study (feasibility phase) will open. Both phases will remain open concurrently and patients will be able to enroll on the Phase 0 then "roll over" and enroll on the feasibility phase. During the feasibility phase patients will be administered tocilizumab every two weeks for up to 13 cycles (approximately 1 year). Patients will be followed for up to 5 years in the feasibility phase.

ELIGIBILITY:
Inclusion Criteria

Phase 0 Eligibility:

1. Tumor biopsy/resection and/or cyst aspiration planned for the clinical care of the patient independent of study participation by the treating pediatric neurosurgeon and neuro-oncologist
2. Must meet one of the following criteria:

   1. Presumed craniopharyngioma based on imaging features and best judgement of treating medical team (if newly diagnosed)
   2. Previous histologically confirmed ACP that has progressed or recurred at the time of enrollment

Feasibility Eligibility:

1. Must meet one of the following criteria:

   1. Recurrent or progressive* ACP treated with surgery alone without radiation
   2. Recurrent or progressive* ACP treated with surgery and radiation

      * Progressive disease for eligibility purposes will be defined as follows: Solid disease: any growth deemed progression based on discretion of the investigator regardless of timing from RT Cystic disease: must be at least 6 months from last day of RT. Patients demonstrating isolated cyst growth >6 months after RT must show a continued increase in the cystic component on two serial MRI scans performed at least 4 weeks apart OR at least partial reaccumulation of the cyst following one or more cyst aspirations.
   3. Newly diagnosed, by histology or imaging ACP with unresectable residual cystic and/or solid disease that is measurable in 2 dimensions
2. Subjects who participated in the Phase 0 portion and meet eligibility, may enroll in the Feasibility Phase of the study once open.

Overall Study Inclusion Criteria:

1. Age: ≥ 2 years and < 21 years
2. Subjects may have received prior tocilizumab or other IL6 or IL6R inhibitor
3. Organ Function Requirements

   1. Adequate bone marrow function defined as:

      * Platelet count ≥100,000/μl (transfusion independent)
      * Absolute neutrophil count (ANC) ≥1500/μl
   2. Adequate renal function defined as:

      * Creatinine clearance or radioisotope GFR ≥70 ml/min/1.73 m2 or
      * A serum creatinine based on age/gender as follows: (Age, Male, Female) 3 to < 6 years, 0.8, 0.8; 6 to < 10 years, 1, 1; 10 to < 13 years, 1.2, 1.2; 13 to < 16 years, 1.5, 1.4; 16 years to < 18 years, 1.7, 1.4
   3. Adequate liver function defined as:

      * SGOT (AST) and SGPT (ALT) <1.5x ULN for age
4. Subjects must meet one of the following performance scores:

   1. ECOG performance status scores of 0, 1, or 2;
   2. Karnofsky score of ≥60 for patients > 16 years of age; or
   3. Lansky score of ≥60 for patients ≤16 years of age
5. Subjects of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
6. Informed consent and assent obtained as appropriate.

Exclusion Criteria

1. Pregnant or breastfeeding
2. Uncontrolled intercurrent illness including, but not limited to:

   1. ongoing or active infection (including active tuberculosis)
   2. symptomatic congestive heart failure
   3. unstable angina pectoris
   4. cardiac arrhythmia
   5. psychiatric illness/social situations that would limit compliance with study requirements are not eligible.
3. Known hypersensitivity or history of anaphylaxis to tocilizumab
4. Received any live vaccinations within 3 months prior to start of therapy
5. Evidence of metastatic disease or other cancer
6. Inability to return for follow up visits or obtain required follow-up studies to assess toxicity of therapy

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 0: Presence of Tocilizumab and Metabolites | Within 4 to 8 hours of administration of tocilizumab
  Utilize biopsy and/or drainage to identify the presence of tocilizumab and its metabolites in adamantinomatous craniopharyngioma (ACP) tumor tissue and/or cyst fluid and/or CSF following one dose of systemically administered tocilizumab.
Feasibility Phase: Toxicity Profile | Start of study to end of study, up to 5 years
  To define toxicities of tocilizumab therapy using CTCAE version 5.

SECONDARY OUTCOMES:
Phase 0: IL6 and Inflammatory Cytokines | Within 4 to 8 hours of administration of tocilizumab
  To define levels of IL6 and other inflammatory cytokines in biopsied tissue and/or cyst fluid as measured by enzyme-linked immunosorbent assay (ELISA) following 1 dose of systemically administered tocilizumab
Feasibility Phase: Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Utilize radiography to estimate PFS of subjects with newly diagnosed, unresectable or recurrent/progressive ACP (with or without prior radiation therapy) treated with systemic tocilizumab.
Feasibility Phase: Pathway Activation | Start of study to end of study, up to 5 years
  To demonstrate evidence of WNT (Wingless-related integration site) in tumor tissue using immunohistochemistry and transcription array
Feasibility Phase: Pathway Activation | Start of study to end of study, up to 5 years
  To demonstrate evidence of MAPK (mitogen activated protein kinases) in tumor tissue using immunohistochemistry and transcription arr
Feasibility Phase: Immunity | Start of study to end of study, up to 5 years
  To demonstrate immune cell infiltration in tumor tissue using immunohistochemistry and flow cytometry
Feasibility Phase: Cytokines | Start of study to end of study, up to 5 years
  To characterize cytokine signaling in tumor tissue and/or cyst fluid using enzyme-linked immunosorbent assay (ELISA)To characterize cytokine signaling in tumor tissue and/or cyst fluid using enzyme-linked immunosorbent assay (ELISA)
Feasibility Phase: Overall Response Rate (ORR) | Start of study to end of study, or up to 5 years
  Utilize radiography to estimate the overall response rate of subjects with newly diagnosed, unresectable or recurrent/progressive ACP (with or without prior radiation therapy) treated with systemic tocilizumab.
Feasibility Phase: 1-Year Disease Stabilization | Start of study to 1 year post treatment
  Utilize radiography to estimate the 1-year disease stabilization rate of subjects with newly diagnosed, unresectable or recurrent/progressive ACP (with or without prior radiation therapy) treated with systemic tocilizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Macy, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No